CLINICAL TRIAL: NCT01773616
Title: Phase 3 Open Label Randomised Multicentre Controlled Trial of Rituxmab and Mycophenolate Mofetil Without Oral Steroids for the Treatment of Lupus Nephritis
Brief Title: Trial of Rituximab and Mycophenolate Mofetil Without Oral Steroids for Lupus Nephritis
Acronym: RITUXILUP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study assessments for patients recruited continuing per protocol so patients receive a minimum of 6 months follow up. No safety concerns have been raised.
Sponsor: Imperial College London (Other)
Collaborators: Karolinska Institutet (Other); Ohio State University (Other); Dutch Working Party on Systemic Lupus Erythematosus (Unknown); EULAR Lupus Nephritis Trial Network Study Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRO2035
Record Dates: First submitted 2012-11-01; First posted 2013-01-23 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Systemic Lupus Erythematosus, Lupus Nephritis
Keywords: Systemic lupus erythematosus; Lupus; Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Nephritis | interventions — Prednisolone; Rituximab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Rituximab, methyl prednisolone and mycophenolate mofetil
  Interventions: Drug: Rituximab; Drug: Mycophenolate mofetil; Drug: Methyl prednisolone
- Oral prednisolone (Active Comparator): Oral prednisolone, methyl prednisolone and mycophenolate mofetil
  Interventions: Drug: Oral prednisolone; Drug: Mycophenolate mofetil; Drug: Methyl prednisolone

INTERVENTIONS:
Drug: Oral prednisolone
  Arms: Oral prednisolone
Drug: Rituximab
  Other Names: MabThera
  Arms: Rituximab
Drug: Mycophenolate mofetil
  Other Names: Cellcept; Myfenax
Drug: Methyl prednisolone

SUMMARY:
The treatment of the multisystem autoimmune disease systemic lupus erythematosus (SLE) remains a challenge, particularly when there is renal involvement (lupus nephritis). For the last 60 years corticosteroids have been the backbone of the treatment of lupus nephritis but they are associated with significant toxicity.

Although randomized placebo controlled trials of Rituximab in non-renal lupus and lupus nephritis did not meet their primary end-points, there is accumulating data that suggests that B cell depletion with Rituximab may be efficacious in lupus disease refractory to conventional therapy. Furthermore, our pilot data suggests that the addition of Rituximab to mycophenolate mofetil (MMF) without oral steroids is at least as effective at inducing a renal response as the standard of care therapy comprising MMF and high dose oral corticosteroids.

RITUXILUP is a proof of concept, open labeled, randomized, controlled, multicentre trial that aims to demonstrate whether the addition of Rituximab to MMF therapy is useful in treating a new flare of lupus nephritis and whether it has a long lasting steroid-sparing, beneficial effect with equal efficacy and greater safety than a conventional regimen of MMF and oral prednisolone. If successful, this trial has the potential to dramatically change the management of lupus nephritis.

DETAILED DESCRIPTION:
TRIAL SUMMARY

TITLE RITUXILUP - An open label randomised multicentre controlled trial of RITUXImab and mycophenolate mofetil (MMF) without oral steroids for the treatment of LUPus nephritis

OBJECTIVES

1. Is the combination of Rituximab, Methyl prednisolone and MMF as effective in treating lupus nephritis as Methyl prednisolone, oral steroids and MMF?
2. Does the omission of oral steroids increase the safety of the treatment regimen?

DESIGN This is a 1:1 randomised, international open label, controlled phase III multicentre trial

SAMPLE SIZE A total of 252 patients: 126 patients in each arm (As of April 2017 decided 25 patients will be maximum recruited following decision to close the study early)

ELIGIBILITY Children (12 years and above) and adults with lupus nephritis ISN/RPS Class III A or A/C, Class IV-G A or A/C, Class IV-S A or A/C, and/or Class V with a urine protein/creatinine ratio (PCR) ≥ 100mg/mmol.

TREATMENT

1. Experimental group - Rituximab, IV methyl prednisolone and mycophenolate mofetil
2. Control group - oral prednisolone, IV methyl prednisolone and mycophenolate mofetil.

PRIMARY OUTCOME The primary outcome is to demonstrate non-inferiority of the Rituximab arm in comparison to the control arm in the proportion of patients achieving complete renal response (CR) at week 52 without the need for steroid prescription.

SECONDARY OUTCOMES

Safety outcomes:

* Serious Infectious Episodes
* Serious Adverse Events
* Evidence of metabolic abnormalities particularly new onset diabetes

Disease control over time:

* Proportion of patients achieving Partial Response (PR)
* Time to stable CR
* Time to PR
* Proportion of patients in PR who achieve histological remission in those who have a repeat biopsy as part of local standard of care
* Proportion of patients with renal or extra flare
* Cumulative steroid exposure
* Deviation from the steroid taper in the steroid arm and/or introduction of steroids in the steroid-free arm
* Proportion of patients achieving a response as defined by the SLE Responder Index (SRI) at week 52 and annually thereafter as defined by:

  * a >4 point reduction in SELENA-SLEDAI score;
  * no new BILAG A organ domain score;
  * no more than I new BILAG B score;
  * no worsening in physician's global assessment (PGA) by >10%;
  * must not have received non-protocol treatment.
* Proportion of patients achieving a response as defined by the BILAG-based Composite Lupus Assessment (BICLA) at week 52 and annually thereafter as defined by: BILAG-2004 improvement (BILAG A to B/C/D, BILAG B to C/D and no BILAG worsening, no deterioration in SLEDAI total score, no worsening in physician's global assessment (PGA) by >10% and must not have received non-protocol treatment.

ELIGIBILITY:
1. Adults aged 18-75 years old and children aged 12-17 years old.
2. Active lupus nephritis, as defined by kidney biopsy within prior 8 weeks assessed by the International Society of Nephrology/Renal Pathology Society (ISN/RPS) classification:

   1. class III (A or A/C) with active lesions in at least 20% of the viable glomeruli, or
   2. class IV-S (A or A/C) with active lesions in at least 20% of the viable glomeruli, or
   3. class IV-G (A or A/C) with active lesions in at least 20% of the viable glomeruli and / or
   4. class V and
   5. urine protein-to-creatinine ratio equal to or greater than 100mg/mmol (>1mg/mg ) at randomisation or at any time within 28 days before randomisation
3. No contraindications to the use of IV methyl prednisolone, MMF, oral steroids or rituximab or any other required medications such as antipyretics, antihistamines
4. Ability to provide informed consent
5. As MMF is teratogenic and on basis of advice from NHS England (The updated recommendations (https://www.gov.uk/drug-safety-update/mycophenolate-mofetil-mycophenolic-acid-new-pregnancy-prevention-advice-for-women-and-men) for patients whilst on MMF and after stopping are:

   * Women who have child bearing potential should be willing to use 2 forms of effective contraception during treatment and for 6 weeks after stopping treatment
   * Men (including those who have had a vasectomy) should be willing to use condoms during treatment and for at least 90 days after stopping treatment. This advice is a precautionary measure due to the genotoxicity of these products
   * Female partners of male patients treated with mycophenolate mofetil should use highly effective contraception during treatment and for 90 days after the last dose

Exclusion criteria:

1. Obsolescence of >50% of the glomeruli or tubulointerstitial scarring of >50% or cellular crescents in >50% of the glomeruli
2. Severe "critical" SLE flare defined as:

   1. BILAG 2004 A flare in CNS system
   2. or any SLE manifestation requiring more immunosuppression than allowed within the protocol in the physician's opinion
3. Pregnant or lactating. Woman who have child bearing potential must have two negative pregnancy test results with a sensitivity of ≥ 25 mIU/mL: one from a serum pregnancy test at day -8 to day -10 of screening and another from a urine pregnancy test at day 1 prior to randomisation. If the timeline is shortened because of clinical urgency, then there must be a negative serum pregnancy test with a sensitivity of ≥ 25 mIU/mL within 1-2 days before study start
4. Patients not willing for their GP to be informed of their participation in this study
5. Patients should not be on or require maintenance steroids and should not have had more than 12 weeks of steroids in the period immediately preceding recruitment irrespective of dose
6. Patients that had received more than 2.0g of IV methyl prednisolone in the previous 4 weeks
7. Prior use within 12 months of screening visit of therapeutic monoclonal antibody, or B or T cell modulating 'biologic' use
8. Prior use within 6 months of the screening visit of Intravenous immunoglobulin / plasma exchange OR Cyclophosphamide
9. Active infections, including but not limited to the human immunodeficiency virus (HIV), and hepatitis B (including prior infection as judged by positive Hepatitis B core antibody) or Hepatitis C or tuberculosis
10. Receipt of a live-attenuated vaccine within 3 months of study enrolment
11. In the investigator's opinion, patients that are at high risk for infection (including but not limited to indwelling catheter, dysphagia with aspiration, decubitus ulcer, history of prior aspiration pneumonia or recurrent severe urinary tract infection)
12. Prior history of invasive fungal infections
13. History of any cancer
14. In female patients, known history of cervical dysplasia CIN Grade III cervical high risk human papillomavirus or abnormal cervical cytology other than abnormal squamous cells of undetermined significance (ASCUS) within the past 3 years. The patient will be eligible after the condition has resolved (e.g., follow-up HPV test is negative or cervical abnormality has been effectively treated >1 year ago)
15. Any concomitant medical condition or abnormal blood results that in the investigator's opinion, or after discussion with the CI, places the participant at risk by participating in this study.
16. Comorbidities requiring systemic corticosteroid therapy.
17. Current substance abuse.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Complete renal response (CR) at week 52 without the need to prescribe oral steroids within 1 year | 1 year
  The proportion of participants who achieve a complete renal response at week 52 without the need to prescribe oral steroids within 1 year, except for one course of maximum 30mg for a maximum of 14 days OR one intramuscular or intra-articular injection of steroids

SECONDARY OUTCOMES:
Serious Infectious Episodes, Serious Adverse Events and Adverse events | 2 years
  4. Metabolic abnormalities related to steroid exposure: 5. Cumulative steroid exposure over 1 and 2 years 6. Introduction of oral steroids in the B cell depleted patients 7. Patients requiring >10mg oral prednisolone at 1 year and 2 year
Metabolic abnormalities related to steroid exposure | 2 years
Cumulative steroid exposure over 1 and 2 years | 2 years
Introduction of oral steroids in the B cell depleted patients | 2 years
Patients requiring >10mg oral prednisolone at 1 year and 2 year | 2 years
Proportion of patients achieving CR at 6, 18 and 24 months | 2 years
Proportion of patients achieving PR at 6,12,8 and 24 months | 2 years
  PR is defined as:
  i) eGFR at baseline or <20% decrease, ii) AND if not nephrotic at baseline (PCR<300mg/mmol), 50% improvement in urine PCR iii) OR if nephrotic at baseline (PCR >300mg/mmol), 50% improvement in urine PCR AND PCR <300mg/mmol
Mean time to stable CR and mean time to PR | 2 years
Proportion of patients in PR who achieve histological remission as judged by absence of proliferative lesions and no new subendothelial or subepithelial deposits | 2 years
Proportion of patients with only 1 or fewer BILAG 2004 Bs in any non-renal organ system at 1 year | 2 years
Proportion of patients with renal flare | 2 years
  Flare is identified by:
  i) Proteinuria >50% increase ii) AND above 100mg/mmol for 2 visits iii) and / or in those with normal renal function and normal urinary sediment, a fall of >20% in eGFR on 2 occasions Where possible flare should be proven by repeat renal biopsy.
Mean time to renal flare in patients achieving CR and PR | 2 years
Proportion of patients achieving normal serum C3,C4 and anti-dsDNA antibodies at week 52 | 2 years

OTHER OUTCOMES:
Patients requiring repeat dosing with Rituximab | 2 years
Patients requiring the addition of any new cytotoxic | 2 years
Patients with non-renal BILAG 2004 A scores or flare and time to A flare | 2 years
Improvement in LupusQoL©, SF-36, EQ5D between baseline, 1 year, 2, 3 and 4 years | 2 years
Patients achieving therapeutic drug levels as a measure of adherence - as judged by mycophenolic acid and hydroxychloroquine levels | 2 years
Relationship between completeness and duration of B cell depletion and achievement of primary end point | 2 years
Patients with decreased immunoglobulin levels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Liz Lightstone, Dr, Study Director — Imperial College London
Locations (11):
- United Kingdom (11):
  - Queen Elizabeth Hospital, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Chapel Allerton Hospital, The Leeds Teaching Hospitals NHS Trust, Leeds
  - Leicester General Hospital, University Hospitals of Leicester NHS Trust, Leicester
  - Royal Free London NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - King's College Hospital, London
  - Manchester Royal Infirmary, Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Churchill Hospital, Oxford University Hospitals NHS Trust, Oxford
  - Royal Stoke Hospital, University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

REFERENCES:
- [Background] If Rituximab together with MMF is shown to be as good as standard treatment with MMF and oral steroids, it would be the first time in 60 years that patients with lupus nephritis could be spared the burden of long term steroids.
- See also: Related Info — http://www1.imperial.ac.uk/clinicaltrialsunit/currenttrials/